CLINICAL TRIAL: NCT04990388
Title: A Phase 1/2 First-in-human, Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses and Repeat Doses of UX053 in Patients With GSD III
Brief Title: Safety, Tolerability, and Pharmacokinetics of UX053 in Patients With Glycogen Storage Disease Type III (GSD III)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision not related to safety concerns
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UX053-CL101; 2021-000903-19 (EudraCT Number)
Record Dates: First submitted 2021-07-26; First posted 2021-08-04 (Actual); Results first posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Glycogen Storage Disease Type III
MeSH Terms: conditions — Glycogen Storage Disease Type III | interventions — Antipyretics; Acetaminophen; Ibuprofen; Histamine H2 Antagonists; Famotidine; Histamine Antagonists; Cetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The SAD and OL-RD cohorts will be open-label, while the DB-RD dose cohorts will be randomized, double-blind, and placebo-controlled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- UX053 Dose Level 1S ->OL-1R (Experimental): Participants receive a single, peripheral intravenous (IV) infusion of UX053. After completion of the 90-day Follow up Period, participants can enter the open label repeat dose (OL-RD) cohort where they will receive UX053 every 4 weeks (Q4W) for 4 doses. Participants will also receive premedication, consisting of oral paracetamol/acetaminophen or ibuprofen, an H2 blocker, and an H1 blocker.
  Interventions: Biological: UX053; Drug: Antipyretic; Drug: H2 Blocker; Drug: H1 Blocker
- UX053 Dose Level 2S->OL-2R (Experimental): Participants receive a single, peripheral intravenous (IV) infusion of UX053. After completion of the 90-day Follow up Period, participants can enter the open label repeat dose (OL-RD) cohort where they will receive UX053 every 4 weeks (Q4W) for 4 doses. Participants will also receive premedication, consisting of oral paracetamol/acetaminophen or ibuprofen, an H2 blocker, and an H1 blocker.
  Interventions: Biological: UX053; Drug: Antipyretic; Drug: H2 Blocker; Drug: H1 Blocker
- UX053 Dose Level 3S->OL-3R (Experimental): Participants receive a single, peripheral intravenous (IV) infusion of UX053. After completion of the 90-day Follow up Period, participants can enter the open label repeat dose (OL-RD) cohort where they will receive UX053 every 4 weeks (Q4W) for 4 doses. Participants will also receive premedication, consisting of oral paracetamol/acetaminophen or ibuprofen, an H2 blocker, and an H1 blocker.
  Interventions: Biological: UX053; Drug: Antipyretic; Drug: H2 Blocker; Drug: H1 Blocker
- UX053 or Placebo Dose Level DB-1R (Experimental): Participants randomized to receive a single, peripheral IV infusion of UX053 or Placebo every 2 weeks (Q2W) for 5 doses. Participants will also receive premedication, consisting of oral paracetamol/acetaminophen or ibuprofen, an H2 blocker, and an H1 blocker.
  Interventions: Biological: UX053; Other: Placebo; Drug: Antipyretic; Drug: H2 Blocker; Drug: H1 Blocker
- UX053 Dose Level DB-2R (Experimental): Participants randomized to receive a single, peripheral IV infusion of UX053 or Placebo every 2 weeks (Q2W) for 5 doses. Participants will also receive premedication, consisting of oral paracetamol/acetaminophen or ibuprofen, an H2 blocker, and an H1 blocker.
  Interventions: Biological: UX053; Other: Placebo; Drug: Antipyretic; Drug: H2 Blocker; Drug: H1 Blocker
- UX053 Dose Level DB-3R (Experimental): Participants randomized to receive a single, peripheral IV infusion of UX053 or Placebo every 2 weeks (Q2W) for 5 doses. Participants will also receive premedication, consisting of oral paracetamol/acetaminophen or ibuprofen, an H2 blocker, and an H1 blocker.
  Interventions: Biological: UX053; Other: Placebo; Drug: Antipyretic; Drug: H2 Blocker; Drug: H1 Blocker

INTERVENTIONS:
Biological: UX053 — mRNA-based biologic
Other: Placebo — consists of the same components as the formulation buffer for UX053
  Arms: UX053 Dose Level DB-2R; UX053 Dose Level DB-3R; UX053 or Placebo Dose Level DB-1R
Drug: Antipyretic — participants will receive oral premedication prior to infusion
  Other Names: paracetamol; acetaminophen; ibuprofen
Drug: H2 Blocker — participants will receive oral premedication prior to infusion
  Other Names: famotidine
Drug: H1 Blocker — participants will receive oral premedication prior to infusion
  Other Names: cetirizine

SUMMARY:
The primary objective of the study is to evaluate the safety of UX053 in adults with Glycogen Storage Disease Type III (GSD III).

DETAILED DESCRIPTION:
This study is a phase 1/2 first-in-human (FIH), study to evaluate the safety, tolerability, and pharmacokinetic (PK) of a single ascending dose (SAD) and repeat doses (RD) of UX053 in patients with GSD III. The SAD cohorts will be open-label (OL). There will be two types of RD cohorts, an open-label (OL-RD) and a randomized, double-blind (DB), and placebo-controlled (DB-RD).

ELIGIBILITY:
Key Inclusion Criteria:

* Confirmed diagnosis of GSD III by gene sequencing or enzymatic testing
* Alanine aminotransferase at or below 5 times normal during the three months prior to dosing
* Willing and able to comply with standard dietary management of GSD III

Inclusion Criteria for Participants Rescreening Into OL-RD Cohorts After Treatment with UX053 in SAD Cohort:

* If a significant rise in ALT occurs after the prior dose, ALT should show a decreasing trend toward the subject's baseline value
* Total bilirubin, platelets and international normalized ratio (INR) is within normal limits

Key Exclusion Criteria:

* History of liver transplant or currently awaiting liver transplant
* History of cirrhosis
* Active Hepatitis B or C
* Severe kidney impairment
* History of liver cancer or large liver tumors
* History of any cancer within the past 3 years
* Known history of HIV infection
* Known severe allergy to polyethylene glycol (PEG), polysorbate, or mRNA vaccine
* Heart failure that causes marked limitation in physical activity
* Poorly controlled diabetes
* Poorly controlled hypothyroidism
* Treatment with immunosuppressive medications such as those used to treat chronic autoimmune conditions and solid organ transplants
* Pregnant or nursing, or planning to become pregnant during the study

Exclusion Criteria for Participants Rescreening Into OL-RD Cohorts After Treatment with UX053 in SAD Cohort:

* New or worsening symptoms of liver disease (including new or worsening hepatomegaly) along with any increase in transaminase levels
* Receipt of any blood product administration (eg, packed red blood cells, platelet, FFP) for management of consumptive coagulopathy
* An ALT level that is ≥ 8x ULN and > 2x the participants baseline value in the absence of an alternative explanation

Note: Additional inclusion/exclusion criteria may apply, per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (6):
- United States (4):
  - University of California, Irvine, Orange, California
  - Rare Disease Research, Atlanta, Georgia
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Texas, Health Science Center of Houston, Houston, Texas
- Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico, Milan, Italy
- Hospital Universitario 12 de Octubre, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ultragenyx Patient Advocacy/GSD III Disease Information — https://ultrarareadvocacy.com/glycogen-storage-disease-type-iii-gsdiii/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 9 participants enrolled in this study; 1 withdrew consent prior to group assignment, did not receive study drug, and was not included in any data table. Eight participants enrolled and were treated; all completed participation in the single ascending dose (SAD) cohorts and were included in the final analysis. None of these participants were randomized, as they were only in SAD cohorts, and none rolled into an open label-repeated dose cohort, as the study discontinued early.
Groups:
- SAD Cohort 1: 0.05 mg/kg: Participants received a single, peripheral intravenous (IV) infusion of a 0.05 mg/kg dose of UX053.
- SAD Cohort 2: 0.10 mg/kg: Participants received a single, peripheral IV infusion of a 0.10 mg/kg dose of UX053.
Period: Overall Study
Arm/Group | SAD Cohort 1: 0.05 mg/kg | SAD Cohort 2: 0.10 mg/kg
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SAD Cohort 1: 0.05 mg/kg | SAD Cohort 2: 0.10 mg/kg | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.20 (5.21) | 43.53 (10.10) | 47.86 (8.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 4 | 7
  Black or African American | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, Deaths, Discontinuations, and/or Dose Changes
Description: An AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. A TEAE is defined as any AE not present prior to the initiation of the drug treatment or any AE already present that worsens in either intensity or frequency following exposure to the drug treatment. An SAE is an AE that meets any of the following criteria in the view of either the Investigator or Ultragenyx: death; life-threatening; inpatient hospitalization or prolongation of existing hospitalization; disability/Incapacity; congenital anomaly/birth defect not present at screening; other important medical events. Severity of events were graded as mild (grade1), moderate (grade 2), severe (grade 3), life-threatening (grade 4), or death (grade 5).
Time Frame: From first dose of study drug through the end of study (up to Day 90)
Measure: Count of Participants; unit: Participants
Arm/Group | SAD Cohort 1: 0.05 mg/kg | SAD Cohort 2: 0.10 mg/kg
Number analyzed (Participants) | 4 | 4
Participants
  Any TEAE | 3 | 4
  Serious TEAE | 0 | 0
  Related TEAE | 0 | 1
  Serious Related TEAE | 0 | 0
  TEAE With Maximum Severity Grade 5 | 0 | 0
  TEAE With Maximum Severity Grade 4 | 0 | 0
  TEAE With Maximum Severity Grade 3 | 0 | 0
  TEAE With Maximum Severity Grade 2 | 0 | 0
  TEAE With Maximum Severity Grade 1 | 3 | 4
  TEAE Leading to Study Discontinuation | 0 | 0
  TEAE Leading to Treatment Discontinuation | 0 | 0
  TEAE Leading to Death | 0 | 0
  TEAE Leading to Dose Reduction | 0 | 0
  TEAE Leading to Dose Interruption | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK) of Amylo-α-1,6-glucosidase 4-alpha-glucanotransferase Messenger Ribonucleic Acid (AGL mRNA) and the Excipient ATX95: Maximum Blood/Plasma Concentration (Cmax)
Time Frame: Pre-infusion; 1, 3, 4, 4.5, 5 hr (± 10 min), 6 hr (± 20 min), 8, 10 hr (± 30 min), 24 hr (± 2 hr), 96, 168 hr (± 24 hr), 336, 504, 672 hr (± 48 hr) post-start of infusion
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SAD Cohort 1: 0.05 mg/kg | SAD Cohort 2: 0.10 mg/kg
Number analyzed (Participants) | 4 | 4
ng/mL
  AGL mRNA | 56.00 (30.59) | 72.15 (60.99)
  ATX95 | 7010.00 (1360.71) | 8585.00 (4439.62)

3. Secondary Outcome: PK of AGL mRNA and the Excipient ATX95: Time to Peak Drug Concentration (Tmax)
Time Frame: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | SAD Cohort 1: 0.05 mg/kg | SAD Cohort 2: 0.10 mg/kg
Number analyzed (Participants) | 4 | 4
hours
  AGL mRNA | 6.10 [4.5 to 7.9] | 6.15 [2.8 to 8.1]
  ATX95 | 4.20 [3.0 to 4.4] | 3.90 [3.0 to 4.1]

4. Secondary Outcome: PK of AGL mRNA and the Excipient ATX95: Total Drug Exposure to the Last Measurable Concentration (AUC0-last)
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | SAD Cohort 1: 0.05 mg/kg | SAD Cohort 2: 0.10 mg/kg
Number analyzed (Participants) | 4 | 4
ng*h/mL
  AGL mRNA | 2567.5 (956.4) | 3931.0 (4191.2)
  ATX95 | 25350.0 (3087.1) | 31350.0 (20738.8)

5. Secondary Outcome: PK of AGL mRNA and the Excipient ATX95: Total Drug Exposure to Infinity (AUC0-inf)
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | SAD Cohort 1: 0.05 mg/kg | SAD Cohort 2: 0.10 mg/kg
Number analyzed (Participants) | 4 | 4
ng*h/mL
  AGL mRNA | 2572.5 (958.0) | 3948.5 (4178.7)
  ATX95 | 25375.0 (3055.5) | 31425.0 (20758.0)

6. Secondary Outcome: PK of AGL mRNA and the Excipient ATX95: Elimination Half-life (t½)
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | SAD Cohort 1: 0.05 mg/kg | SAD Cohort 2: 0.10 mg/kg
Number analyzed (Participants) | 4 | 4
hours
  AGL mRNA | 53.8 (4.3) | 44.8 (11.6)
  ATX95 | 18.0 (7.5) | 32.3 (32.2)

7. Secondary Outcome: PK of AGL mRNA and the Excipient ATX95: Clearance (CL)
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/h/kg
Arm/Group | SAD Cohort 1: 0.05 mg/kg | SAD Cohort 2: 0.10 mg/kg
Number analyzed (Participants) | 4 | 4
mL/h/kg
  AGL mRNA | 21.42 (7.16) | 55.51 (52.36)
  ATX95 | 39.80 (4.62) | 94.73 (69.18)

8. Secondary Outcome: PK of AGL mRNA and the Excipient ATX95: Volume of Distribution at Steady State (Vss)
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | SAD Cohort 1: 0.05 mg/kg | SAD Cohort 2: 0.10 mg/kg
Number analyzed (Participants) | 4 | 4
mL/kg
  AGL mRNA | 1638.8 (722.4) | 3993.3 (3546.5)
  ATX95 | 167.8 (76.0) | 741.5 (874.0)

ADVERSE EVENTS:
Time Frame: Up to 90 days after dosing.
Groups:
- Total: Participants received a single, peripheral IV infusion of a 0.05 or 0.10 mg/kg dose of UX053.
Arm/Group | SAD Cohort 1: 0.05 mg/kg | SAD Cohort 2: 0.10 mg/kg | Total
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/8
Other Adverse Events (participants affected / at risk) | 3/4 | 4/4 | 7/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SAD Cohort 1: 0.05 mg/kg (N=4) | SAD Cohort 2: 0.10 mg/kg (N=4) | Total (N=8)
Pyrexia (General disorders) | 1 | 0 | 1
Seasonal Allergy (Immune system disorders) | 1 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Joint Injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Haematoma (Vascular disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1
Ear infection bacterial (Infections and infestations) | 1 | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/88/NCT04990388/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT04990388/SAP_001.pdf